CLINICAL TRIAL: NCT01314755
Title: A Double Blind, Randomised, Placebo Controlled, Feasibility Phase III Clinical Trial of Peri-operative Immune-enhancing Feed in Patients Undergoing Surgery for Advanced Head and Neck Cancer
Brief Title: A Trial of Perioperative Immune Enhancing Feed in Patients Undergoing Surgery for Head and Neck Cancer
Acronym: IMPACTHN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terrence Jones (Other Government)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor-Investigator, Terrence Jones, Professor, Liverpool University Hospitals NHS Foundation Trust
Organization: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC.73.03
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Squamous Cell Carcinoma of Mouth; Squamous Cell Carcinoma of Oropharynx; Laryngeal Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Hypopharynx
Keywords: Head and Neck neoplasm; Nutrition; Carcinoma; Infection; Post-operative; Surgery; Immune-enhancing
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma; Infections

STUDY DESIGN:
Intervention Model Description: either Impact or an iso-nitrogenous, iso-caloric control feed for five days pre and seven days post-surgery
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- immune-enhancing feed IMPACT (Experimental): immune-enhancing feed IMPACT
  Interventions: Dietary Supplement: IMPACT
- control arm (Active Comparator): iso-nitrogenous, iso-caloric control feed
  Interventions: Dietary Supplement: An iso-caloric, iso-nitrogenous control feed

INTERVENTIONS:
Dietary Supplement: IMPACT — IMPACT (Nestlé Healthcare Nutrition, Minnetonka, MN, USA) an 'immune-enhancing' feed which contains supplemental L-arginine (1.25 78 g/L), dietary nucleotides (1.2 g/L) and omega-3 fatty acids in the form of 79 eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) (EPA/DHA 1.7 g/L) 80 as its active ingredients.
  Arms: immune-enhancing feed IMPACT
Dietary Supplement: An iso-caloric, iso-nitrogenous control feed
  Arms: control arm

SUMMARY:
Study Hypothesis: The peri-operative enteral administration of a proprietary immune-enhancing feed (IMPACT) will not reduce post-operative infective complications in patients undergoing major surgery for squamous cell carcinoma of the Head and neck (SCCHN).

Patients who present with SCCHN for whom surgery is the recommended treatment will, assuming they fulfill the eligibility criteria, be block randomised into a two-group, double-blind randomised controlled trial. One group will receive IMPACT, the other an iso-caloric, iso-nitrogenous control feed for 5 days pre and 7 days post-operatively. In both groups patients will be fed enterally. The feeds will be prepared in identical bottles to facilitate blinding. Primary outcome measures include major systemic infection, whilst secondary outcome measures include local infection and length of hospital stay. Follow-up will be for 30 days postsurgery.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

Patients who were to undergo either of the following procedures

* partial (external approach) or total laryngectomy
* partial pharyngectomy with primary closure or free-flap reconstruction
* total pharyngectomy (gastric (or colonic) transposition, other free flap reconstruction, or other pedicled flap reconstruction)
* oral cavity or oropharyngeal resection requiring reconstruction with a free flap or pedicled flap

Exclusion Criteria:

Patients with

* malabsorption syndromes
* primary immune disorders
* active infection on presentation
* patients undergoing secondary surgical reconstruction
* patients undergoing palliative surgery
* patients aged under 18 years old
* patients who were pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2003-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Systemic infection | 30 days post surgery
  Lower respiratory tract; Gastro-intestinal tract; Urinary tract; Haematological.

SECONDARY OUTCOMES:
Local/wound site infection | Within 30 days post-surgery
  Local/wound site infection
Length of post-operative hospital stay | Up to 30 days post surgery
  Length of post-operative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Terence M Jones, MD, Principal Investigator — University of Liverpool
Locations (1):
- University Hospital Aintree, Liverpool, Merseyside, United Kingdom